CLINICAL TRIAL: NCT05852717
Title: A Phase II Trial Evaluating Safety and Efficacy of Epcoritamab With Gemcitabine, Dexamethasone, and Cisplatin (GDP) Salvage Chemotherapy in Relapsed Refractory Large B-cell Lymphoma
Brief Title: Safety and Efficacy of Epcoritamab With Gemcitabine, Dexamethasone, and Cisplatin (GDP) Salvage Chemotherapy in Relapsed Refractory Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dipenkumar Modi (Other)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor-Investigator, Dipenkumar Modi, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LYM22-565
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Large Cell Lymphoma, Diffuse; Relapsed Cancer; Refractory Cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Neoplasms | interventions — Immunotherapy, Adoptive; Transplantation, Autologous; Receptors, Chimeric Antigen; Automobiles; Guanosine Diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GDP + Epcoritamab + AutoSCT or CAR T-cell therapy (Experimental): Cycles 1-3 (Cycle = 21 days) Epcoritamab will be administered by subcutaneous injection Days 1, 8, and 15. Epcoritamab Day 1: 0.16mg, Day 8: 0.8mg, Day 15: 48mg except Cycle 2-Epcoritamab will administered at 48mg on Days 1, 8 and 15
  Gemcitabine will be administered by IV infusion on Days 1 and 8. Gemcitabine Days 1,8: 1,000mg/m^2
  Cisplatin will be administered by IV infusion on Day 1. Cisplatin Day 1: 75mg/m^2
  Dexamethasone will be given by mouth on Days 1-4. Dexamethasone Days 1-4: 40mg
  After completion of Cycle 3 Autologous stem cell transplant (AutoSCT) OR CAR T-cell therapy
  Interventions: Procedure: AutoSCT OR CAR T-cell Therapy; Drug: GDP; Drug: Epcoritamab
- GDP + Epcoritamab + Epcoritamab Maintenance (Experimental): Cycles 1-3 (Cycle = 21 days) Epcoritamab will be administered by subcutaneous injection Days 1, 8, and 15 of each Cycle.
  Epcoritamab Day 1: 0.16mg, Day 8: 0.8mg, Day 15: 48mg except Cycle 2-Epcoritabab will administered at 48mg on Days 1, 8 and 15
  Gemcitabine will be administered by IV infusion on Days 1 and 8 of each Cycle. Gemcitabine Days 1,8: 1,000mg/m^2
  Cisplatin will be administered by IV infusion on Day 1 of each Cycle. Cisplatin Day 1: 75mg/m^2
  Dexamethasone will be given by mouth on Days 1-4 of Cycle 1 ONLY. Dexamethasone Days 1-4: 40mg
  Cycles 4-9 (Cycle =28 Days) Epcoritamab will be administered by subcutaneous injection on Days 1, 8, and 15 of Cycles 4-9.
  Interventions: Drug: GDP; Drug: Epcoritamab

INTERVENTIONS:
Procedure: AutoSCT OR CAR T-cell Therapy — Autologous stem cell transplant (AutoSCT) or CAR T-cell therapy will be performed after Cycle 3 of receiving epcoritamab and GDP
  Other Names: Autologous transplant; chimeric antigen receptor (CAR) T-cell
  Arms: GDP + Epcoritamab + AutoSCT or CAR T-cell therapy
Drug: GDP — Gemcitabine Cisplatin Dexamethasone
Drug: Epcoritamab — Epcoritamab

SUMMARY:
Subjects with relapsed large cell lymphoma will receive 3 cycles of combination therapy consisting of GDP and epcoritamab. Each cycle will last 21 days. GDP consists of gemcitabine 1000 mg/m2 IV on Days 1 and 8, cisplatin 75 mg/m2 IV on Day 1, and dexamethasone 40 mg orally on Days 1 through 4. Epcoritamab will be administered subcutaneously (SC) on Days 1, 8, and 15. Patients will receive granulocyte colony stimulating factor (G-CSF) between Day 8 through Day 10 of each cycle of combination therapy.

Patients will then undergo radiology imaging for disease assessment. Patients may proceed to SCT(autologous or allogeneic) or CAR T-cell therapy or epcoritamab monotherapy upon completion of Cycle 3 per investigator discretion. The rationale for subjects not proceeding to autoSCT or CAR T-cell therapy will be captured in the eCRFs.

Patients who do not undergo SCT or CAR T-cell therapy may have the option to receive study treatment with epcoritamab monotherapy following completion of Cycle 3. Epcoritamab monotherapy will be offered to selected subjects who become ineligible to undergo SCT or CAR T-cell therapy (such as social situation, change in subject decision). The decision to offer epcoritamab monotherapy will be per investigator's discretion. However, subjects must have demonstrated a response to the combination therapy (partial remission or complete remission) per disease assessment scans prior to offering epcoritamab monotherapy. Epcoritamab monotherapy should begin 2 weeks following Cycle 3 Day 15. Monotherapy will consist of epcoritamab 48 mg administered subcutaneously on Days 1 and 15 of each 28 day cycle for Cycle 4 to Cycle 9 or until unacceptable toxicity, or disease progression per the Lugano Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-2 within 28 days prior to registration.
4. Histologically confirmed CD20+ relapsed large cell lymphoma according to the 5th edition of the WHO classification of the hematolymphoid tumors and the 2022 international consensus classification of mature lymphoid neoplasms. This includes de-novo and transformed from prior indolent B-cell NHL such as follicular lymphoma, or marginal zone lymphoma (33, 34). Subjects with high-grade B-cell lymphoma (HGBCL), NOS subtype, and high-grade B-cell lymphoma with c-MYC, Bcl2 and/or Bcl6 rearrangements (double or triple hit lymphoma) are eligible. Patients with primary mediastinal B-cell lymphoma, and T-cell histiocyte-rich B-cell lymphoma, primary cutaneous diffuse large B-cell lymphoma, leg type, Intravascular large B-cell lymphoma, Epstein-Barr virus-positive diffuse large B-cell lymphoma, NOS, Diffuse large B-cell lymphoma associated with chronic inflammation, and ALK-positive large B-cell lymphoma are eligible. Patients with Burkitt lymphoma or lymphoplasmacytic lymphoma are not eligible.
5. Positron emission tomography (PET) positive measurable disease with at least 1 node having the longest diameter (LDi) greater than (>) 1.5 centimeter (cm) or 1 extranodal lesion with LDi >1 cm (per the Lugano Criteria 2014).
6. Have received at least 1 prior line of systemic therapy for the treatment of large cell lymphoma. NOTE: Prior radiation therapy or systemic corticosteroids will not be considered a line of therapy.
7. Patients must be deemed eligible to proceed with stem cell transplantation (autologous or allogeneic) or CAR T-cell therapy per treating physician discretion. Patients being considered for allogeneic stem cell transplant may be eligible. Patients with prior stem cell transplantation or CAR T-cell therapy are eligible if they are deemed eligible to undergo another stem cell transplantation or CAR T-cell therapy.
8. Must have had relapsed or refractory disease following standard frontline chemotherapy. Refractory disease is defined as large cell lymphoma not achieving complete remission, progressing, or relapsing within 6 months after first-line chemotherapy based on PET/CT per the Lugano criteria. Relapsed disease is defined as disease that recurs beyond 6 months after completion of initial chemotherapy based on PET/CT per the Lugano criteria.
9. Archival tissue obtained within 2 years of signing consent is required if available and will be identified at screening and shipped prior to Cycle 2 Day 1. If archival tissue is not available, but the subject is undergoing a standard of care biopsy, fresh tissue from that standard of care biopsy may be used for eligibility. If a subject does not have archival tissue obtained within 2 years of signing consent or is not undergoing a standard of care biopsy, they are not eligible for the trial. Cytological or fine-needle aspiration samples are not acceptable. Tumor tissue from bone metastases that has been decalcified is not acceptable.
10. Demonstrate adequate organ function. All screening labs to be obtained within 21 days prior to registration. *Patients with bone marrow involvement will be eligible to participate in the study but must meet hematologic parameters.
11. Life expectancy of ≥ 6 months, as determined by the enrolling physician or protocol designee.
12. Females subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study treatment. If a urine test is done and it is positice ir cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential and male subjects must be willing to abstain from penile-vaginal intercourse or to use an effective method(s) of contraception.
14. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Previous treatment with gemcitabine, cisplatin, and epcoritamab or other bispecific T-cell engager antibody (BsAB) such as glofitamab, mosunetuzumab, or odronextamab.
2. Known active central nervous system or meningeal involvement by large cell lymphoma at time of screening. Patients diagnosed with CNS disease who achieved and maintained CNS CR at the time of relapse are eligible. Lumbar puncture must be done in this case prior to study entry to demonstrate CNS CR status. Tests to investigate CNS involvement are required otherwise only if clinically indicated (i.e. disease suspected on basis of symptoms or other findings).
3. Contraindication to any drug contained in the combination therapy regimen (GDP).
4. Known hypersensitivity or allergic reaction to epcoritamab or its' excipients.
5. Use of any standard or experimental anti-large cell lymphoma therapy (including nonpalliative radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy) < 14 days prior to C1D1. NOTE: Prednisone up to 50 mg or equivalent for 5 days is permitted; palliative radiation is permitted only if on non-target lesions).
6. Major surgery < 14 days of Cycle 1 Day 1.
7. Neuropathy Grade ≥ 2 (CTCAE v.5.0).
8. Patients with a history of other malignancies, except adequately treated non-melanoma skin cancer, non-invasive superficial bladder cancer, curatively treated in-situ cancer of the cervix, DCIS of the breast, localized low grade prostate cancer (up to Gleason score 6), or other solid tumours curatively treated with no evidence of disease for at least 3 years.
9. Active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) requiring systemic treatment within 7 days prior to the first dose of study treatment. Prophylactic antibacterial, antiviral, and antifungal agents are allowed.
10. Active HIV infection. NOTE: Testing for HIV antibody is required at the time of screening. Those with positive HIV antibody will require HIV viral load by PCR testing. Patients with detectable viral load will not be eligible for the study. Those with positive antibody but undetectable viral load and CD4 >200 will be eligible.
11. Testing for hepatitis B (HBV) and hepatitis C virus (HCV) is required at screening. Hepatitis B testing will consist of Hepatitis B surface Antigen (HBsAg), Hepatitis B Core Antibody (HBcAb) and Hepatitis Surface Antibody (HBsAb). Hepatitis C testing will consist of Hepatitis C Antibody (HCAb). Subjects with a history of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated. Subjects with evidence of prior HBV but who are PCR-negative are permitted in the trial but should receive prophylactic antiviral therapy. Subjects with a history of hepatitis C virus (HCV) infection must have been treated. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. Subjects who received treatment for HCV that was intended to eradicate the virus may participate if hepatitis C RNA levels are undetectable.
12. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
13. Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety, or being compliant with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | 4 years
  CR rate is defined as proportion of subjects with a CR based on the Lugano Criteria 2022 following 3 cycles of combination treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 4 years
  ORR is defined as the proportion of subjects with a CR + PR based on Lugano Criteria 2022
Duration of Response (DOR) | 4 years
  DOR is defined as time from first observed response (CR or PR) to date of progression (PD) based on the Lugano Criteria 2022 or death, whichever occurs first.
Progression-free Survival (PFS) | 4 years
  PFS is defined as the time from treatment initiation until disease progression based on the Lugano Criteria 2022 or death from any cause.
Overall Survival (OS) | 4 years
  OS is defined as the time from treatment initiation until death from any cause.
Feasibility of AutoSCT or CAR T-cell | 6 months
  Feasibility of stem cell mobilization or CAR T-cell therapy will be assessed based on the number of subjects that undergo autologous transplant or CAR T-cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dipenkumar Modi, MD, Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Karmanos Cancer Center (Wayne State University), Detroit, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia